CLINICAL TRIAL: NCT00496314
Title: Clinical Study Assessing Physician's Comfort Level and Satisfaction When Using The e2TM Cervical Cell Collector Compared to the Standard Spatula/CytoBrush Technique
Brief Title: Physician's Comfort Level and Satisfaction Study With The e2TM Collector Compared to the Spatula/CytoBrush Technique
Status: Terminated | Type: Observational
Why Stopped: Terminated for lack of resources to complete.
Sponsor: CytoCore, Inc. (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Other Study IDs: 12-20-06
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Cervical Cell Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: e2TM Cervical Cell Collector

SUMMARY:
A study which assesses the physician's comfort level and satisfaction when using the e2TM Collector compared to the Spatula/SytoBrush technique.

ELIGIBILITY:
Inclusion Criteria:

* Every Physician who will participate in the two CytoCore prospective studies assessing the safety and efficacy of the e2TM Collector
* Each physician will have used the Collector 15 - 25 times
* Each physician will have signed the Consent form prior to using the Collector for the first time.

Exclusion Criteria:

* None (commensurate with the above inclusion conditions.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Physician comfort level and satisfaction when using the e2TM Collector compared to the standard spatula/cytobrush. | Each physician will be surveyed after first and last use of the e2TM collector as well as three more times spaced at near regular intervals in between.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pinkerton, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospital CASE Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Sankaranarayanan R, Budukh AM, Rajkumar R. Effective screening programmes for cervical cancer in low- and middle-income developing countries. Bull World Health Organ. 2001;79(10):954-62. Epub 2001 Nov 1. PMID 11693978
- [Background] Umland B, Waterman R, Wiese W, Duban S, Mennin S, Kaufman A. Learning from a rural physician program in China. Acad Med. 1992 May;67(5):307-9. doi: 10.1097/00001888-199205000-00004. No abstract available. PMID 1575861
- [Background] Holowaty P, Miller AB, Rohan T, To T. RESPONSE: re: natural history of dysplasia of the uterine cervix. J Natl Cancer Inst. 1999 Aug 18;91(16):1420A-1421. doi: 10.1093/jnci/91.16.1420a. No abstract available. PMID 10451450
- [Background] Solomon D, Davey D, Kurman R, Moriarty A, O'Connor D, Prey M, Raab S, Sherman M, Wilbur D, Wright T Jr, Young N; Forum Group Members; Bethesda 2001 Workshop. The 2001 Bethesda System: terminology for reporting results of cervical cytology. JAMA. 2002 Apr 24;287(16):2114-9. doi: 10.1001/jama.287.16.2114. PMID 11966386
- [Background] Nanda K, McCrory DC, Myers ER, Bastian LA, Hasselblad V, Hickey JD, Matchar DB. Accuracy of the Papanicolaou test in screening for and follow-up of cervical cytologic abnormalities: a systematic review. Ann Intern Med. 2000 May 16;132(10):810-9. doi: 10.7326/0003-4819-132-10-200005160-00009. PMID 10819705
- [Background] Fahey MT, Irwig L, Macaskill P. Meta-analysis of Pap test accuracy. Am J Epidemiol. 1995 Apr 1;141(7):680-9. doi: 10.1093/oxfordjournals.aje.a117485. PMID 7702044
- [Background] Clavel C, Masure M, Bory JP, Putaud I, Mangeonjean C, Lorenzato M, Nazeyrollas P, Gabriel R, Quereux C, Birembaut P. Human papillomavirus testing in primary screening for the detection of high-grade cervical lesions: a study of 7932 women. Br J Cancer. 2001 Jun 15;84(12):1616-23. doi: 10.1054/bjoc.2001.1845. PMID 11401314
- [Background] Willis BH, Barton P, Pearmain P, Bryan S, Hyde C. Cervical screening programmes: can automation help? Evidence from systematic reviews, an economic analysis and a simulation modelling exercise applied to the UK. Health Technol Assess. 2005 Mar;9(13):1-207, iii. doi: 10.3310/hta9130. PMID 15774236
- [Background] Buntinx F, Brouwers M. Relation between sampling device and detection of abnormality in cervical smears: a meta-analysis of randomised and quasi-randomised studies. BMJ. 1996 Nov 23;313(7068):1285-90. doi: 10.1136/bmj.313.7068.1285. PMID 8942687
- [Background] Martin-Hirsch P, Lilford R, Jarvis G, Kitchener HC. Efficacy of cervical-smear collection devices: a systematic review and meta-analysis. Lancet. 1999 Nov 20;354(9192):1763-70. doi: 10.1016/s0140-6736(99)02353-3. PMID 10577637
- [Background] Martin-Hirsch P, Jarvis G, Kitchener H, Lilford R. Collection devices for obtaining cervical cytology samples. Cochrane Database Syst Rev. 2000;2000(2):CD001036. doi: 10.1002/14651858.CD001036. PMID 10796736
- [Background] Selvaggi SM, Guidos BJ. Specimen adequacy and the ThinPrep Pap Test: the endocervical component. Diagn Cytopathol. 2000 Jul;23(1):23-6. doi: 10.1002/1097-0339(200007)23:13.0.CO;2-K. PMID 10907927
- [Background] Marchand L, Mundt M, Klein G, Agarwal SC. Optimal collection technique and devices for a quality pap smear. WMJ. 2005 Aug;104(6):51-5. PMID 16218317
- [Background] Koss LG. Evolution in cervical pathology and cytology: a historical perspective. Eur J Gynaecol Oncol. 2000;21(6):550-4. No abstract available. PMID 11214608